CLINICAL TRIAL: NCT04752033
Title: Intrathecal Opioids for Pain Control After Colorectal Resection: Determining the Optimal Dose
Brief Title: Intrathecal Opioids for Colorectal Resection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adam Amundson MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-009205
Record Dates: First submitted 2021-01-28; First posted 2021-02-12 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Surgery; Pain, Postoperative; Analgesic, Opioid
Keywords: Intrathecal; Morphine; Hydromorphone; Dose Finding
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Hydromorphone

STUDY DESIGN:
Intervention Model Description: Dose Finding Study Utilizing Sequential Up and Down Method Using Biased Coin Design
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Morphine (Experimental): Subjected to sequential up and down dose titration using biased coin method in parallel with the hydromorphone arm
  Interventions: Drug: Morphine
- Hydromorphone (Experimental): Subjected to sequential up and down dose titration using biased coin method in parallel with the morphine arm
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Morphine — Dose titration utilizing will be done using sequential up and down design using biased coin method. All participant will receive a morphine dose that is within the range of doses currently utilized clinically and no participant will receive placebo only.
  Arms: Morphine
Drug: Hydromorphone — Dose titration utilizing will be done using sequential up and down design using biased coin method. All participant will receive a hydromorphone dose that is within the range of doses currently utilized clinically and no participant will receive placebo only.
  Arms: Hydromorphone

SUMMARY:
This research study is being done to determine the optimal dose of spinal morphine and hydromorphone in patients undergoing minimally-invasive (i.e., surgery performed through small entry sites and using cameras) colorectal surgery.

DETAILED DESCRIPTION:
Intrathecal (IT) opioids have been established as a safe and efficacious modality to treat postoperative pain. In the setting of colorectal surgery, studies have shown that intrathecal opioids together with multimodal analgesic regimens provide pain relief superior to multimodal analgesia alone. Furthermore, in the setting of multimodal analgesia, IT opioids also appear to be equianalgesic to epidural analgesia while conferring an improved safety profile. As a result, many institutions have incorporated intrathecal opioids into their Enhanced Recovery after Surgery (ERAS) pathways.

While morphine has traditionally been considered the "gold standard" in IT opioid therapy for postsurgical pain, hydromorphone has been gaining popularity as an alternative. The doses ranging between 0.005 mg to 0.25 mg for hydromorphone12-15 and 0.05 mg to 0.625 mg (with doses as high as 10 mcg/kg in the setting of cardiac surgery) for morphine has been found to be efficacious in this patient population. However, increasing opioid doses are associated with increased incidence of adverse effects. A meta-analysis reviewing twenty-eight studies which investigated intrathecal morphine versus placebo demonstrated moderate increases in the incidences of pruritus, nausea and vomiting. In fact, the incidence of nausea with IT morphine has been reported to be 33%. While hydromorphone is similar chemically to morphine, it is metabolized differently. Differences in pharmacokinetics may allow for differences in side effect profiles. Hydromorphone is more lipid soluble than morphine. This decreases its spread within the intrathecal space and enhances its penetration into the dorsal horn of the spinal cord where interactions with opioid receptors occur. Some studies (performed in the women undergoing cesarean delivery) have also found that hydromorphone causes less nausea and pruritus than morphine, while others have not.

Despite the widespread use of IT hydromorphone and morphine for pain after colorectal surgery, the optimal dose for neither drug has been established in prospective trials. The investigators have previously performed a dose-finding study of IT hydromorphone and morphine in women undergoing cesarean delivery. Briefly, 80 parturients scheduled for elective cesarean delivery were randomized to receive IT morphine or IT hydromorphone at a dose determined using up-down sequential allocation with a biased-coin design to determine ED90, which was found to be 75 mcg for IT hydromorphone and 150 mcg for IT morphine. The follow-up study performed by the investigators also found no differences in adverse effects or efficacy between the drugs. The results from the obstetric population, however, cannot be directly translated to the colorectal surgery population due to pharmacodynamic and pharmacokinetics differences related to the pregnancy, age, presence of comorbidities, differences in surgical techniques, and co-administration of IT local anesthetic.

This study applies the methodology the investigators have previously used in the obstetric population to the patients undergoing colorectal resection and aims to identify the optimal dose of IT hydromorphone and morphine that provides good pain relief without causing significant side effects. Secondarily, the investigators will compare each drug at its optimal dose in terms of opioid consumption and side effects. Based on their prior findings, the investigators hypothesize that the optimal dose of intrathecal hydromorphone will be 75 mcg and the optimal dose of intrathecal morphine will be 150 mcg. Additionally, the investigators hypothesize that exploratory findings comparing the two drugs at their optimal doses will show no difference in the incidence of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with an American Society of Anesthesiologists (ASA) physiological status I-III.
* Undergoing colorectal minimally invasive surgery (MIS).
* Age between 18 and 75 years of age.
* Body mass index (BMI) between 18.5 and 40.
* Ability to understand and read English.

Exclusion Criteria:

* Not able or unwilling to sign consent.
* Patients undergoing ileostomy closure.
* Patients undergoing ambulatory surgery or anticipated to be discharged sooner than 24 hours after surgery
* Patients with chronic pain, requiring daily opioid use at the time of surgery.
* Patient intolerant or allergic to opioids, NSAIDs, or acetaminophen.
* Patients requiring emergent surgery.
* Any contraindication to neuraxial anesthesia (coagulopathy, localized infection at the site of injection, pre-existing spinal pathology, or peripheral neuropathy).
* Any patients currently receiving any anticoagulation medication other than aspirin and who have not discontinued the medication per American Society of Regional Anesthesia anticoagulation guidelines22, and/or an abnormal INR.
* Patients with hepatic or renal insufficiency in as much as the patient is not a candidate for acetaminophen or NSAIDs, respectively.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam W Amundson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vinsard PA, Pleticha J, Sharpe EE, Panchamia JK, Olsen DA, Sviggum HP, Shawki SF, Behm KT, Larson DW, LeMahieu AM, Niesen AD, Amundson AW. A Prospective Randomized Dose-Finding Study of Intrathecal Opioids for Postoperative Analgesia After Minimally Invasive Colorectal Operation. Mayo Clin Proc Innov Qual Outcomes. 2025 Mar 3;9(2):100600. doi: 10.1016/j.mayocpiqo.2025.100600. eCollection 2025 Apr. PMID 40114986
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Morphine 50 mcg; Morphine 100 mcg; Morphine 150 mcg; Morphine 200 mcg; Morphine 250 mcg; Morphine 300 mcg; Morphine 350 mcg; Morphine 400 mcg: Subjected to sequential up and down dose titration using biased coin method in parallel with the hydromorphone arm
  Morphine: Dose titration utilizing will be done using sequential up and down design using biased coin method. All participant will receive a morphine dose that is within the range of doses currently utilized clinically and no participant will receive placebo only.
- Hydromorphone 50 mcg; Hydromorphone 75 mcg; Hydromorphone 100 mcg; Hydromorphone 125 mcg; Hydromorphone 150 mcg; Hydromorphone 175 mcg; Hydromorphone 200 mcg: Subjected to sequential up and down dose titration using biased coin method in parallel with the morphine arm
  Hydromorphone: Dose titration utilizing will be done using sequential up and down design using biased coin method. All participant will receive a hydromorphone dose that is within the range of doses currently utilized clinically and no participant will receive placebo only.
Period: Overall Study
Arm/Group | Morphine 50 mcg | Morphine 100 mcg | Morphine 150 mcg | Morphine 200 mcg | Morphine 250 mcg | Morphine 300 mcg | Morphine 350 mcg | Morphine 400 mcg | Hydromorphone 50 mcg | Hydromorphone 75 mcg | Hydromorphone 100 mcg | Hydromorphone 125 mcg | Hydromorphone 150 mcg | Hydromorphone 175 mcg | Hydromorphone 200 mcg
Started | 2 | 5 | 4 | 4 | 4 | 1 | 4 | 16 | 6 | 10 | 6 | 2 | 1 | 3 | 12
Completed | 2 | 5 | 4 | 4 | 4 | 1 | 4 | 16 | 6 | 10 | 6 | 2 | 1 | 3 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Morphine 100 mcg: Subjected to sequential up and down dose titration using biased coin method in parallel with the hydromorphone arm
  Hydromorphone: Dose titration utilizing will be done using sequential up and down design using biased coin method. All participant will receive a hydromorphone dose that is within the range of doses currently utilized clinically and no participant will receive placebo only.
- Morphine 150 mcg; Morphine 200 mcg; Morphine 250 mcg; Morphine 300 mcg; Morphine 350 mcg; Morphine 400 mcg: Subjected to sequential up and down dose titration using biased coin method in parallel with the hydromorphone arm
- Hydromorphone 50 mcg; Hydromorphone 75 mcg; Hydromorphone 100 mcg; Hydromorphone 125 mcg; Hydromorphone 150 mcg; Hydromorphone 175 mcg; Hydromorphone 200 mcg: Subjected to sequential up and down dose titration using biased coin method in parallel with the morphine arm
- Total: Total of all reporting groups
Arm/Group | Morphine 50 mcg | Morphine 100 mcg | Morphine 150 mcg | Morphine 200 mcg | Morphine 250 mcg | Morphine 300 mcg | Morphine 350 mcg | Morphine 400 mcg | Hydromorphone 50 mcg | Hydromorphone 75 mcg | Hydromorphone 100 mcg | Hydromorphone 125 mcg | Hydromorphone 150 mcg | Hydromorphone 175 mcg | Hydromorphone 200 mcg | Total
Number analyzed (Participants) | 2 | 5 | 4 | 4 | 4 | 1 | 4 | 16 | 6 | 10 | 6 | 2 | 1 | 3 | 12 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 4 | 4 | 3 | 1 | 3 | 15 | 4 | 8 | 6 | 0 | 1 | 3 | 8 | 66
  >=65 years | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 0 | 2 | 0 | 0 | 4 | 14
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [27 to 64] | 40 [37 to 73] | 45 [23 to 58] | 47.5 [39 to 64] | 57.5 [44 to 71] | 39 | 56 [46 to 70] | 54 [29 to 71] | 65.6 [36 to 70] | 53 [24 to 68] | 51 [27 to 62] | 73 [73 to 73] | 33 | 44 [20 to 46] | 62 [19 to 71] | 52 [34 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 3 | 2 | 2 | 0 | 3 | 8 | 2 | 4 | 3 | 1 | 0 | 0 | 8 | 41
  Male | 2 | 0 | 1 | 2 | 2 | 1 | 1 | 8 | 4 | 6 | 3 | 1 | 1 | 3 | 4 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 00 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
    White | 2 | 5 | 4 | 3 | 4 | 1 | 4 | 16 | 6 | 9 | 6 | 2 | 1 | 3 | 11 | 77
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 5 | 4 | 4 | 4 | 1 | 4 | 16 | 6 | 10 | 6 | 2 | 1 | 3 | 12 | 80
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 28.9 [27.1 to 30.7] | 26.9 [19.8 to 43.1] | 27.2 [24.8 to 32] | 35.1 [27.4 to 39.2] | 25.75 [22.8 to 31.7] | 27.81 | 24.6 [18.5 to 29.4] | 30.55 [22.6 to 37.4] | 28.4 [18.2 to 31.4] | 28.5 [20 to 40] | 30 [24.2 to 34.4] | 28.95 [26.4 to 31.5] | 21.53 | 29.8 [28.3 to 36.3] | 26.3 [18.5 to 36.2] | 28 [25.2 to 32]

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Control
Description: Failure was reported as a pain score of over 4/10 on a Numeric Rating Scale (NRS), scale range 0-10, 0 being no pain and 10 being the worst pain imaginable
Time Frame: 12 hours after intrathecal (IT) drug administration
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Morphine 50 mcg | Morphine 100 mcg | Morphine 150 mcg | Morphine 200 mcg | Morphine 250 mcg | Morphine 300 mcg | Morphine 350 mcg | Morphine 400 mcg | Hydromorphone 50 mcg | Hydromorphone 75 mcg | Hydromorphone 100 mcg | Hydromorphone 125 mcg | Hydromorphone 150 mcg | Hydromorphone 175 mcg | Hydromorphone 200 mcg
Number analyzed (Participants) | 2 | 5 | 4 | 4 | 4 | 1 | 4 | 16 | 6 | 10 | 6 | 2 | 1 | 3 | 12
score on a scale | 4.5 [2 to 7] | 1.6 [1 to 4] | 1.75 [0 to 4] | 2.75 [1 to 6] | 3.75 [0 to 8] | 8 | 3.75 [2 to 5] | 3.31 [0 to 9] | 3 [0 to 7] | 3.2 [0 to 7] | 1.6 [0 to 3] | 2.5 [2 to 3] | 4 | 4.3 [3 to 5] | 2.5 [1 to 10]

2. Secondary Outcome: Postoperative Pain Control
Description: Reported as Numeric Rating Scale (NRS), scale range 0-10, 0 being no pain and 10 being the worst pain imaginable.
Time Frame: 24 hours after IT drug administration
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Morphine 50 mcg | Morphine 100 mcg | Morphine 150 mcg | Morphine 200 mcg | Morphine 250 mcg | Morphine 300 mcg | Morphine 350 mcg | Morphine 400 mcg | Hydromorphone 50 mcg | Hydromorphone 75 mcg | Hydromorphone 100 mcg | Hydromorphone 125 mcg | Hydromorphone 150 mcg | Hydromorphone 175 mcg | Hydromorphone 200 mcg
Number analyzed (Participants) | 2 | 5 | 4 | 4 | 4 | 1 | 4 | 16 | 6 | 10 | 6 | 2 | 1 | 3 | 12
units on a scale | 3 [2 to 4] | 2.2 [0 to 4] | 2.25 [1 to 4] | 3 [0 to 6] | 4.25 [3 to 7] | 7 | 4.5 [2 to 7] | 3.37 [0 to 8] | 4.33 [2 to 8] | 3.72 [1 to 7] | 2.4 [1 to 4] | 3.5 [3 to 4] | 3 | 3.66 [1 to 7] | 4 [0 to 10]

3. Secondary Outcome: Presence and Severity of Opioid-related Side Effects at Their Highest Doses
Description: Nausea and vomiting, pruritus, sedation, respiratory depression. The ordinal subjective scale of mild, moderate, and severe will be used.
Time Frame: 12 and 24 hours after IT drug administration
Population: At 12 hours and 24 hours
Measure: Number; unit: participants
Groups:
- Hydromorphone 50 mcg; Hydromorphone 75 mcg; Hydromorphone 100 mcg; Hydromorphone 125 mcg; Hydromorphone 150 mcg; Hydromorphone 175 mcg; Hydromorphone 200 mcg: Subjected to sequential up and down dose titration using biased coin method in parallel with the arm morphine
  Hydromorphone: Dose titration utilizing will be done using sequential up and down design using biased coin method. All participant will receive a morphine dose that is within the range of doses currently utilized clinically and no participant will receive placebo only.
Arm/Group | Morphine 50 mcg | Morphine 100 mcg | Morphine 150 mcg | Morphine 200 mcg | Morphine 250 mcg | Morphine 300 mcg | Morphine 350 mcg | Morphine 400 mcg | Hydromorphone 50 mcg | Hydromorphone 75 mcg | Hydromorphone 100 mcg | Hydromorphone 125 mcg | Hydromorphone 150 mcg | Hydromorphone 175 mcg | Hydromorphone 200 mcg
Number analyzed (Participants) | 2 | 5 | 4 | 4 | 4 | 1 | 4 | 16 | 6 | 10 | 6 | 2 | 1 | 3 | 12
participants
  Nausea and Vomiting None at 12 hours | 1 | 2 | 1 | 3 | 0 | 1 | 1 | 7 | 4 | 5 | 2 | 0 | 0 | 1 | 6
  Nausea and Vomiting Mild at 12 hours | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 3 | 2 | 3 | 2 | 1 | 0 | 0 | 3
  Nausea and Vomiting Moderate at 12 hours | 1 | 1 | 1 | 1 | 2 | 0 | 2 | 3 | 0 | 2 | 1 | 1 | 1 | 2 | 1
  Nausea and Vomiting Severe at 12 hours | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Pruritus None at 12 hours | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 0 | 3 | 4 | 1 | 2 | 1 | 0 | 3
  Pruritus Mild at 12 hours | 2 | 1 | 2 | 1 | 2 | 0 | 1 | 5 | 3 | 3 | 3 | 0 | 0 | 2 | 2
  Pruritus Moderate at 12 hours | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 7 | 0 | 2 | 1 | 0 | 0 | 1 | 2
  Pruritus Severe at 12 hours | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 1 | 1 | 0 | 0 | 0 | 5
  Sedation at 12 hours | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory Depression at 12 hours | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea and Vomiting None at 24 hours | 2 | 1 | 3 | 3 | 2 | 1 | 1 | 10 | 6 | 8 | 2 | 2 | 1 | 1 | 7
  Nausea and Vomiting Mild at 24 hours | 0 | 2 | 0 | 1 | 2 | 0 | 3 | 3 | 0 | 2 | 2 | 0 | 0 | 1 | 4
  Nausea and Vomiting Moderate at 24 hours | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
  Nausea and Vomiting Severe at 24 hours | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pruritus None at 24 hours | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 3 | 4 | 0 | 1 | 0 | 0 | 3
  Pruritus Mild at 24 hours | 0 | 2 | 3 | 1 | 3 | 0 | 3 | 5 | 2 | 4 | 3 | 0 | 1 | 0 | 1
  Pruritus Moderate at 24 hours | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 6 | 0 | 1 | 3 | 0 | 0 | 3 | 2
  Pruritus Severe at 24 hours | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 6
  Sedation at 24 hours | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory Depression at 24 hours | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Overall Benefits of Analgesia Score (OBAS)
Description: OBAS is a validated measure incorporating both effectiveness of pain control and unwanted effects related to analgesic treatment. The scale ranges from 0 to 24, with higher the score, worse the pain control.
Time Frame: 12 and 24 hours after highest IT drug administration
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Morphine 50 mcg; Morphine 100 mcg; Morphine 150 mcg; Morphine 200 mcg; Morphine 250 mcg; Morphine 300 mcg; Morphine 350 mcg; Morphine 400 mcg: Subjected to sequential up and down dose titration using biased coin method in parallel with the arm hydromorphone
  Morphine: Dose titration utilizing will be done using sequential up and down design using biased coin method. All participant will receive a morphine dose that is within the range of doses currently utilized clinically and no participant will receive placebo only.
Arm/Group | Morphine 50 mcg | Morphine 100 mcg | Morphine 150 mcg | Morphine 200 mcg | Morphine 250 mcg | Morphine 300 mcg | Morphine 350 mcg | Morphine 400 mcg | Hydromorphone 50 mcg | Hydromorphone 75 mcg | Hydromorphone 100 mcg | Hydromorphone 125 mcg | Hydromorphone 150 mcg | Hydromorphone 175 mcg | Hydromorphone 200 mcg
Number analyzed (Participants) | 2 | 5 | 4 | 4 | 4 | 1 | 4 | 16 | 6 | 10 | 6 | 2 | 1 | 3 | 12
score on a scale
  At 12 hours | 5.5 [2 to 9] | 4.8 [3 to 6] | 2.33 [1 to 4] | 3.5 [1 to 7] | 4.5 [2 to 6] | 3 | 3.33 [1 to 6] | 5.625 [0 to 16] | 2.8 [0 to 8] | 4.09 [2 to 7] | 3 [0 to 5] | 2.5 [1 to 4] | 7 | 5.5 [3 to 8] | 4.5 [0 to 15]
  At 24 hours | 3.5 [0 to 7] | 3.2 [2 to 5] | 2.5 [1 to 4] | 2.75 [2 to 4] | 4 [0 to 10] | 1 | 3.75 [1 to 8] | 5.13 [0 to 16] | 3.6 [0 to 9] | 3.27 [0 to 7] | 3.8 [1 to 6] | 2.5 [2 to 3] | 10 | 4 [0 to 8] | 4.08 [0 to 18]

5. Secondary Outcome: Quality of Recovery (QoR) 15 Score
Description: QoR 15 score is a multidimensional, valid, reliable, responsive, and easy-to-use method of measuring quality in patients' postoperative recovery. The scale ranges from 0 to 150, with higher the score, the better the recovery is.
Time Frame: 24 hours after IT drug administration
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Morphine 50 mcg | Morphine 100 mcg | Morphine 150 mcg | Morphine 200 mcg | Morphine 250 mcg | Morphine 300 mcg | Morphine 350 mcg | Morphine 400 mcg | Hydromorphone 50 mcg | Hydromorphone 75 mcg | Hydromorphone 100 mcg | Hydromorphone 125 mcg | Hydromorphone 150 mcg | Hydromorphone 175 mcg | Hydromorphone 200 mcg
Number analyzed (Participants) | 2 | 5 | 4 | 4 | 4 | 1 | 4 | 16 | 6 | 10 | 6 | 2 | 1 | 3 | 12
score on a scale | 114.5 [98 to 130.5] | 120.5 [105 to 133.5] | 108.5 [90 to 133] | 123.75 [118 to 139] | 106.25 [75 to 139] | 131 | 116.75 [97 to 140] | 115.9 [70 to 142] | 119 [97 to 149] | 119.5 [83 to 135] | 117.8 [105 to 141] | 126 [120 to 132] | 104 | 102 [85 to 125] | 116.75 [39 to 147]

ADVERSE EVENTS:
Time Frame: 12 and 24 hours
Arm/Group | Morphine 50 mcg | Morphine 100 mcg | Morphine 150 mcg | Morphine 200 mcg | Morphine 250 mcg | Morphine 300 mcg | Morphine 350 mcg | Morphine 400 mcg | Hydromorphone 50 mcg | Hydromorphone 75 mcg | Hydromorphone 100 mcg | Hydromorphone 125 mcg | Hydromorphone 150 mcg | Hydromorphone 175 mcg | Hydromorphone 200 mcg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5 | 0/4 | 0/4 | 0/4 | 0/1 | 0/4 | 0/16 | 0/6 | 0/10 | 0/6 | 0/2 | 0/1 | 0/3 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5 | 0/4 | 0/4 | 0/4 | 0/1 | 0/4 | 0/16 | 0/6 | 0/10 | 0/6 | 0/2 | 0/1 | 0/3 | 0/12
Other Adverse Events (participants affected / at risk) | 2/2 | 5/5 | 3/4 | 3/4 | 4/4 | 1/1 | 4/4 | 16/16 | 3/6 | 6/10 | 6/6 | 2/2 | 1/1 | 3/3 | 9/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine 50 mcg (N=2) | Morphine 100 mcg (N=5) | Morphine 150 mcg (N=4) | Morphine 200 mcg (N=4) | Morphine 250 mcg (N=4) | Morphine 300 mcg (N=1) | Morphine 350 mcg (N=4) | Morphine 400 mcg (N=16) | Hydromorphone 50 mcg (N=6) | Hydromorphone 75 mcg (N=10) | Hydromorphone 100 mcg (N=6) | Hydromorphone 125 mcg (N=2) | Hydromorphone 150 mcg (N=1) | Hydromorphone 175 mcg (N=3) | Hydromorphone 200 mcg (N=12)
Nausea and Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) — Mild at 12 hours
Nausea and Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) — Moderate at 12 hours
Nausea and Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Severe at 12 hours
Nausea and Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (4) — Mild at 24 hours
Nausea and Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Moderate at 24 hours
Nausea and Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Severe at 24 hours
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (2) — Mild at 12 hours
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) — Moderate at 12 hours
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) — Severe at 12 hours
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 5 (5) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Mild at 24 hours
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 2 (2) — Moderate at 24 hours
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6) — Severe at 24 hours

LIMITATIONS AND CAVEATS:
Difficulties during patient selection as minimally invasive colorectal surgeries were performed as an outpatient basis negating the use of IT opioids. This issue prolonged patient recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT04752033/Prot_SAP_000.pdf